CLINICAL TRIAL: NCT00266955
Title: A Retrospective Study of Children With ADHD and Cardiac Symptoms
Brief Title: Retrospective of Children With ADHD and Cardiac Symptoms
Status: Terminated | Type: Observational
Why Stopped: insufficient number of eligible subjects
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 04-111
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2007-09

CONDITIONS: Congenital Disorders
Keywords: pediatric; cardiac; ADHD; Adderall; Straterra
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
There is some evidence suggesting ADHD medication interaction could result in mild myocardial ischemia/infarct.

DETAILED DESCRIPTION:
Children with no previous cardiac history who have been on Adderall for ADHD, have developed acute cardiac symptoms after the addition of Straterra for the treatment of ADHD.

We wish to do a study of the medication interactions of Straterra and other ADHD medications focusing on the cardiac manifestations.

We will collect the following information on each patient: Medical Record Number, Account number, Dates of Admission, Discharge, Treatment or Death, Information Regarding Cardiac Signs and Symptoms, Medication Information, Age, Weight, Diagnoses

ELIGIBILITY:
Inclusion Criteria:

* ADHD
* myocardial ischemia/infarct
* no previous cardiac history
* added Straterra
* already taking Adderall

Exclusion Criteria:

* those who do not meet inclusion criteria

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: retro chart review
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 1999-01; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Clabby, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States